CLINICAL TRIAL: NCT00727792
Title: Refinement and Assessment of New MRI Technologies for Thoracic/ Cardiovascular Exams
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Michigan (Other)
Responsible Party: Principal Investigator, Jadranka Stojanovska, M.D., M.S., Principal Investigator, University of Michigan
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: HUM00041514
Record Dates: First submitted 2008-07-28; First posted 2008-08-04 (Estimated); Last update posted 2020-01-21 (Actual); Status verified 2020-01

CONDITIONS: Magnetic Resonance Imaging (MRI) of the Chest
Keywords: participants; scheduled; clinically; ordered; MRI

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Group 2 - Research MRI (Experimental): Subjects will have additional sequences and/or modification to MRI sequences.
  Interventions: Procedure: MRI-Research
- Group 1 - Clinical MRI (Active Comparator): Clinically ordered MRI scan. Subjects will not have any additional sequences or modifications to their clinically ordered MRI
  Interventions: Procedure: MRI -Clinical

INTERVENTIONS:
Procedure: MRI -Clinical — MRI done is standard of care
  Arms: Group 1 - Clinical MRI
Procedure: MRI-Research — MRI includes extra sequences
  Arms: Group 2 - Research MRI

SUMMARY:
The purpose of the study is to improve chest MRI exams, eventually resulting in improvements in patient care.

DETAILED DESCRIPTION:
We will recruit patients to participate in the assessment of new MRI technologies designed to improve chest MRI exams that will result in improvements in patient care.

Several different MRI technologies will be evaluated. Specific evaluation of distinct technologies (eg. new head coil design, and new imaging sequence for the spine) may be evaluated simultaneously, or over non-overlapping periods in time.

ELIGIBILITY:
Inclusion Criteria:

* If you are a male or a non-pregnant female patient, age 18 years or older, of any ethnic background presenting to MRI for a clinically-ordered chest MRI exam, you are eligible to participate in this study.
* If you are a female of child bearing potential you will be questioned for the possibility of pregnancy. Pregnancy screening, if necessary, is performed routinely by ordering physicians prior to MRI scanning to confirm the patient is not pregnant.

Exclusion Criteria:

* Patients who have electrically, magnetically or mechanically activated implants such as heart pacemaker, magnetic surgical clips, prostheses or implanted neurological stimulator.
* Pregnant patients or patients who are nursing
* Patients who are claustrophobic.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2009-01 (Actual); Primary Completion 2019-04-16 (Actual); Study Completion 2019-04-16 (Actual)

PRIMARY OUTCOMES:
New MRI Technologies | 3 years
  Assessment of the new technologies will be quantified by a variety of performance and image quality/content measures. The appropriate set of measures will be selected based on specific features offered by each assessed technology, but will be drawn from the following quantities:
  1. Scan speed: Scan speed is time required to set-up and run the new technique relative to the standard method.
  2. Signal to noise: SNR (signal to noise ratio)is the ratio of average image intensity in target tissue relative to standard deviation of background areas (outside of body). This is a fundamental parameter used to quantify relative performance of new imaging sequences/hardware/software.
  3. Contrast to noise: CNR (contrast to noise)is the difference in average image intensity between two target tissues relative to noise. This is a key descriptor to quantity lesion/tissue conspicuity, thus is used to characterize relative performance of new imaging sequence/hardware/software.

CONTACTS AND LOCATIONS:
Overall Officials: Jadranka Stojanovska, MD, Principal Investigator — University of Michigan
Locations (1):
- University of Michigan Hospital, Ann Arbor, Michigan, United States

IPD SHARING:
Plan to Share IPD: No